CLINICAL TRIAL: NCT07047651
Title: The Effectiveness and Efficacy of the Combination of Pharmacotherapy With the Two New Recovery-oriented Programs, RECOVERYTRSGR (Treatment Resistant Schizophrenia) and RECOVERYTRSBDGR (Treatment Resistant Bipolar Disorder)
Brief Title: Τhe Combination of Pharmacotherapy With RECOVERYTRSGR and RECOVERYTRSBDGR.
Acronym: RAKGEORREC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Stavroula Rakitzi (Other)
Responsible Party: Sponsor-Investigator, Dr. Stavroula Rakitzi, Director, Rakitzi, Stavroula
Organization: Rakitzi, Stavroula (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAKITZI & GEORGILA RECOVERY
Record Dates: First submitted 2025-04-11; First posted 2025-07-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Treatment Resistant Schizophrenia; Treatment Resistant Bipolar Disorder
Keywords: RECOVERYTRSGR; RECOVERYTRSBDGR; Treatment resistant schizophrenia; Treatment resistant bipolar disorder; Recovery-oriented therapy
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Clozapine; Olanzapine; Aripiprazole; Risperidone; asenapine; Paliperidone Palmitate; Clopenthixol; Drug Therapy; Clonazepam; oxybutynin; Antidepressive Agents; Psychotherapy; Lithium; Valproic Acid; Citalopram

STUDY DESIGN:
Intervention Model Description: Pharmacotherapy and RECOVERYTRSGR (190 sessions) will be compared to treatment as usual (TAU) and pharmacotherapy (190 sessions) and Pharmacotherapy and RECOVERYTRSBDGR (140 sessions) will be compared also to TAU and pharmacotherapy (140 sessions).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Pharmacotherapy and RECOVERYTRSGR 22 participants
  Interventions: Combination Product: Group A: (Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol,anxiolytics: clonazepam, stedon, tavor antidepressants: seropram),
- Group B (Active Comparator): Pharmacotherapy and TAU. 20 participants
  Interventions: Combination Product: Group B (Pharmacotherapy and TAU) (Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, antidepressants,
- Group C (Experimental): Pharmacotherapy and RECOVERYTRSBDGR. 22 participants
  Interventions: Combination Product: Group C (Pharmacotherapy and Psychotherapy) Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, lithium, depakine
- Group D (Active Comparator): Pharmacotherapy and TAU. 20 participants
  Interventions: Combination Product: Group D (Pharmacotherapy and TAU)Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, seropram, lithium, depakine)

INTERVENTIONS:
Combination Product: Group A: (Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol,anxiolytics: clonazepam, stedon, tavor antidepressants: seropram), — A combination of pharmacotherapy (antipsychotics, anxiolytics, antidepressants) with RECOVERYTRSGR (psychotherapy) for patients with treatment-resistant schizophrenia. 190 sessions. 22 patients
  Arms: Group A
Combination Product: Group B (Pharmacotherapy and TAU) (Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, antidepressants, — The combination of pharmacotherapy (antipsychotics, anxiolytics, antidepressants) and TAU (psychotherapy) for patients with treatment-resistant schizophrenia. 190 sessions. The control group of Group A 20 patients
  Arms: Group B
Combination Product: Group C (Pharmacotherapy and Psychotherapy) Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, lithium, depakine — A combination of pharmacotherapy with RECOVERYTRSBDGR (antipsychotics, anxiolytics, antidepressants, mood stabilizers) for patients with treatment-resistant bipolar disorder. 140 sessions, 22 people
  Arms: Group C
Combination Product: Group D (Pharmacotherapy and TAU)Clozapine, quietiapine, olanzapine, aripiprazole, zyprasidone, risperidone, asenapine, paliperidone, clopixol, clonazepam, stedon, tavor, seropram, lithium, depakine) — A combination of pharmacotherapy (antipsychotics, anxiolytics, antidepressants, mood stabilizers) and TAU (psychotherapy). A control group to RECOVERYTRSBDGR. 140 sessions. 20 people
  Arms: Group D

SUMMARY:
The effectiveness and efficacy of the combination of pharmacotherapy with the two new recovery-oriented programs, RECOVERYTRSGR for patients with treatment- resistant schizophrenia and RECOVERYTRSBDGR for patients with treatment- resistant bipolar disorder.

DETAILED DESCRIPTION:
RECOVERYTRSGR is a newly developed program for patients with treatment resistant schizophrenia by Dr. S. Rakitzi and Dr. P. Georgila. RECOVERYTRSBDGR is a newly developed program for patients with treatment resistant bipolar disorder by Dr. S. Rakitzi and Dr. P. Georgila. These programs offer a long term combination of pharmacotherapy and cognitive behavioral psychotherapy and rehabilitation and aim to imrove cognition, symptoms, functional outcomes and recovery.

Treatment resistant schizophrenia and treatment resistant bipolar disorder are the most difficult chronic mental health disorders which need long-term treatment.

ELIGIBILITY:
Inclusion Criteria: For patients with treatment resistant schizophrenia:

* age 18-65
* IQ ≥ 80
* Diagnosis TRS.

Inclusion criteria for patients with treatment resistant bipolar disorder:

* age 18-65
* IQ ≥ 80
* Diagnosis TRSBD.

Exclusion Criteria: For patients with treatment resistant schizophrenia:

* Substance abuse and head injury. If substance abuse is successfully treated, the participant will be accepted into our program.
* Relapse and hospitalization.

Exclusion criteria for patients with treatment resistant bipolar diosrder:

* Substance abuse and head injuries. If substance abuse is successfully treated, the participant will be acknowledged into our program.
* Relapse and hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
MCCB BACS symbol coding (for RECOVERYTRSGR) | Pre-intervention
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB BACS symbol coding (for RECOVERYTRSGR) | Immediately after the intervention
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB BACS symbol coding (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB Wechsler memory scale-spatial span (for RECOVERYTRSGR) | Pre-intervention
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better, Summary of forward and backward total score.
MCCB Wechsler memory scale-spatial span (for RECOVERYTRSGR) | Immediately after the intervention
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better. Summary of forward and backward total score
MCCB Wechsler memory scale-spatial span (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better. Summary of forward and backward total score
MCCB Neurospychological Assessment Battery (NAB) (for RECOVERYTRSGR) | Pre-intervention
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Neurospychological Assessment Battery (NAB) (for RECOVERYTRSGR) | Immediately after the intervention
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Neurospychological Assessment Battery (NAB) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Brief visuospatial memory test (for RECOVERYTRSGR) | Pre-intervention
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better.
MCCB Brief visuospatial memory test (for RECOVERYTRSGR) | Immediately after the intervention
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better.
MCCB Brief visuospatial memory test (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Stimuli (for RECOVERYTRSGR) | Pre-intervention
  It measures social cognition. Minimum 0, maximum 67. high scores better.
Social Perception Scale (SPS) Stimuli (for RECOVERYTRSGR) | Immediately after the intervention
  It measures social cognition. Minimum 0, maximum 67. high scores better.
Social Perception Scale (SPS) Stimuli (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures social cognition. Minimum 0, maximum 67. high scores better.
Social Perception Scale (SPS) Interpretation (for RECOVERYTRSGR) | Pre-intervention
  It measures social cognition. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Interpretation (for RECOVERYTRSGR) | Immediately after the intervention
  It measures social cognition. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Interpretation (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures social cognition. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Title (for RECOVERYTRSGR) | Pre-intervention
  It measures social cognition. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Title (for RECOVERYTRSGR) | Immediately after the intervention
  It measures social cognition. Minimum 0, maximum 12. high scores better.
Social Perception Scale (SPS) Title (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures social cognition. Minimum 0, maximum 12. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Pre-intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Pre-intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Immediately after the intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Pre-intervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Pre-intervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Immediately after the intervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Pre-intervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Pre-intervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Immediately after the intervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test (Kosmidou & Vlahou, 2010) (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
PANNS total (for RECOVERYTRSGR) | Pre-intervention
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
PANNS total (for RECOVERYTRSGR) | Immediately after the intervention
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
PANNS total (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
WHODAS total (for RECOVERYTRSGR) | Pre-intervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total (for RECOVERYTRSGR) | Immediately after the intervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
RAS-DS total (for RECOVERYTRSGR) | Pre-intervention
  It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total (for RECOVERYTRSGR) | Immediately after the intervention
  It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures recovery. Minimum 0, maximum 152. High scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Pre-intervention
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Immediately after the intervention
  It. measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It. measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Pre-intervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Immediately after the intervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSGR) | Follow-up up to 24 weeks
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
SRSDA (for RECOVERYTRSBDGR) | Pre-intervention
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA (for RECOVERYTRSBDGR) | Pre-intervention
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
SRSDA (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
SRSDA (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
Hamilton Depression Scale (for RECOVERYTRSBDGR) | Pre-intervention
  It measures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale (for RECOVERYTRSBDGR) | Immediately after the intervention
  It meaasures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It meaasures depression. Minimum 0, maximum 23. Low scores better.
Montgomery and Asperg depression scale (for RECOVERYTRSBDGR) | Pre-intervention
  It measures depression. Minimum 0, maximum 60. Low scores better.
Montgomery and Asperg depression scale (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures depression. Minimum 0, maximum 60. Low scores better.
Montgomery and Asperg depression scale (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures depression. Minimum 0, maximum 60. Low scores better.
The Altman self-rating scale (for RECOVERYTRSBDGR) | Pre-intervention
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
The Altman self-rating scale (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
The Altman self-rating scale (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Pre-intervention
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 44. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 24. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 24. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Pre-intervention
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 44. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 44. Low scores better.
PSYRAT (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 24. Low scores better.
WHODAS total (for RECOVERYTRSBDGR) | Pre-intervention
  It measures functional outcome. Minimum 0, maximum 100. Low scores better.
WHODAS total (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures functional outcome. Minimum 0, maximum 100. Low scores better.
WHODAS total (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures functional outcome. Minimum 0, maximum 100. Low scores better.
RAS-DS Total (for RECOVERYTRSBDGR) | Pre-intervention
  It measures recovery. Minimum 0, maximum 152. High scores better
RAS-DS Total (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures recovery. Minimum 0, maximum 152. High scores better
RAS-DS Total (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures recovery. Minimum 0, maximum 152. High scores better
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Pre-intervention
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Pre-intervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Young mania rating scale (for RECOVERYTRSBDGR) | Pre-intervention
  It measures mania. Minimum 0, maximum 60. Low scores better
The Young mania rating scale (for RECOVERYTRSBDGR) | Immediately after the intervention
  It measures mania. Minimum 0, maximum 60. Low scores better
The Young mania rating scale (for RECOVERYTRSBDGR) | Follow-up up to 24 weeks
  It measures mania. Minimum 0, maximum 60. Low scores better

SECONDARY OUTCOMES:
WAIS (for RECOVERYTRSGR) | Pre-intervention
  It measures the Intelligenz-quotient
WAIS (for RECOVERYTRSBDGR) | Pre-intervention
  It measures the Intelligenz-quotient

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stavroula Rakitzi, PhD, Study Director — Private Practice; Dr. Polyxeni Georgila, M. D., Study Director — Private Practice
Locations (1):
- Private practice of Dr. S. Rakitzi and Dr. P. Georgila ILISION 34 15771 ATHENS GREECE, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
This is the first study regarding the efficacy and effectiveness of RECOVERYTRSGR, and RECOVERYTRSBDGR, which are developed by us.

REFERENCES:
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982
- [Background] 2. Aster, M., Neubauer, M., & Horn R. (2006) Wechsler-Intelligenztest für Erwachsene WIE. Frankfurt: Harcourt Test Services.
- [Background] 3. Bech, P. (1993). Rating scales for Psychopathology, Health Status and Quality of Life. Berlin, Heidelberg, New York: Springer-Verlag.
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] 5. Donias, S., Karastergiou, A., & Manos N. (1991). Standardization of the symptom checklist-90-R rating scale in a Greek population. Psychiatriki, 2(1), 42-48.
- [Background] Fountoulakis KN, Iacovides A, Kleanthous S, Samolis S, Gougoulias K, St Kaprinis G, Bech P. The Greek translation of the symptoms rating scale for depression and anxiety: preliminary results of the validation study. BMC Psychiatry. 2003 Dec 10;3:21. doi: 10.1186/1471-244X-3-21. PMID 14667249
- [Background] 7. Guy, W. (ed). (1976). ECDEU Assessment. Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration, 1976.
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] 9. Hancock, N., Scanlan, J.N., Bundy, A.C., Honey, A. (2019). Recovery Assessment Scale -Domains & Stages (RAS-DS) Manual- Version 3. Sydney: University of Sydney.
- [Background] 10. Hancock, N., & the University of Sydney (2023). Rakitzi S. Katoudi S. Recovery Assessment Scale-Domains & Stages (RAS-DS). The Greek version.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] 12. Kosmidou, M., & Vlahou, Ch. (2010). The Greek verbal memory test. Athens: Parisianos.
- [Background] 13. Koumpouros, Y., Papageorgiou, E., & Sakellari E. et al. (2018). Adaptation and psychometric properties evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. Health Services and Outcomes Research Methodology, 18(1), 63-74. https://doi.org/10.1007/s10742-017-0176-x
- [Background] 14. Lykouras, L., Botsis, A., & Oulis P. (2005). The PANSS Scale. Athens: Scientific Publications.
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] 16. Nuechterlein, K.H., & Green, M.F. (2006). Matrics Consensus Cognitive Battery. MATRICS. Los Angeles: MATRICS Assessment Inc.
- [Background] 17. Rakitzi, S., & Georgila, P. (2024). Treatment resistant schizophrenia. Evidence-based pharmacotherapy, cognitive behavioral psychotherapy and rehabilitation. Springer.
- [Background] 18. Rakitzi, S., & Georgila, P. (2024b). Treatment resistant bipolar disorder. Evidence-based pharmacotherapy, cognitive behavioral psychotherapy and rehabilitation. Springer.
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] 20. World Health Organization. International classification of functioning, disability and health (ICF). Geneva: World Health Organization; 2001.
- [Background] Fuentes, I., Garcia, S., Ruiz, J.C., Soler, J., & Roder, V. (2007). Social perception scale in Schizophrenia. A pilot study. International Journal of Psychology and Psychological therapy, 7 (1), 1-12

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07047651/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07047651/ICF_001.pdf